CLINICAL TRIAL: NCT05341089
Title: A Phase 1 Multiple-Dose Study to Investigate the Pharmacokinetics, Safety, and Tolerability of 2 Different Formulations of LY3502970 in Healthy Participants
Brief Title: A Study of Two Different Formulations of LY3502970 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 17785; J2A-MC-GZGH (Other: Eli Lilly and Company)
Record Dates: First submitted 2022-04-18; First posted 2022-04-22 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09-15

CONDITIONS: Healthy
MeSH Terms: interventions — orforglipron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3502970 (Formulation 1) (Experimental): LY3502970 administered orally.
  Interventions: Drug: LY3502970
- LY3502970 (Formulation 2) (Experimental): LY3502970 administered orally.
  Interventions: Drug: LY3502970

INTERVENTIONS:
Drug: LY3502970 — Administered orally.

SUMMARY:
The main purpose of this study is to conduct blood tests to measure how much LY3502970 is in the bloodstream when administered as two different formulations in healthy participants. The study will also evaluate the safety and tolerability of LY3502970. The study will last up to 13 weeks excluding the screening period.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy as determined by medical evaluation
* Participants who have a hemoglobin level of at least 11.4 grams per deciliter (g/dL) for female participants and at least 12.5 g/dL for male participants
* Participants with a body weight of at least 45 kilograms (kg) and body mass index (BMI) of 18.5 to 35.0 kilograms per meter squared (kg/m²)
* Male participants who agree to use highly effective/effective methods of contraception and female participants not of childbearing potential

Exclusion Criteria:

* Participants who have any abnormality in the 12-lead electrocardiogram (ECG) at screening
* Participants who have an abnormal blood pressure, pulse rate, or both, which are deemed to be clinically significant by the investigator, at screening
* Participants who have known allergies to LY3502970, related compounds, or any components of the formulation
* Participants who have used or intend to use over-the-counter or prescription medication including herbal medications or traditional medications within 14 days prior to dosing
* Participants who show evidence of human immunodeficiency virus (HIV) infection and/or positive HIV antibodies, or both. A negative test within 6 months of screening would not need to be repeated.
* Participants who show evidence of hepatitis C and/or positive hepatitis C antibody, or both. A negative test within 6 months of screening would not need to be repeated.
* Participants who show evidence of hepatitis B, positive hepatitis B surface antigen, and/or positive hepatitis B core antibody, or all. A negative test within 6 months of screening would not need to be repeated.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of LY3502970 | Pre-dose on Day 1 up to 39 days post-dose
  PK: Cmax of LY3502970
PK: Area Under the Plasma Concentration-Time Curve from 0 to 24 hours (AUC0-24) of LY3502970 | Pre-dose on Day 1 up to 39 days post-dose
  PK: AUC0-24 of LY3502970
PK: Time to Maximum Observed Concentration (Tmax) of LY3502970 | Pre-dose on Day 1 up to 39 days post-dose
  PK: Tmax of LY3502970

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Lilly Centre for Clinical Pharmacology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No